CLINICAL TRIAL: NCT01801748
Title: The Natural History of Wheat Hypersensitivity in Thai Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: National Research Council of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 490/2555(EC3)
Record Dates: First submitted 2013-02-26; First posted 2013-03-01 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Wheat Allergy; Child
Keywords: wheat allergy; wheat outgrowing; wheat hypersensitivity; omega-5-gliadin; natural history of wheat hypersensitivity
MeSH Terms: conditions — Wheat Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- oral wheat challenge (Experimental)
  Interventions: Dietary Supplement: oral wheat challenge

INTERVENTIONS:
Dietary Supplement: oral wheat challenge

SUMMARY:
Wheat allergy is affected 0.4-1% and is a major staple of the worldwide diet. Wheat avoidance is exceedingly difficult and imposes major dietary restriction. The purpose of this study were to determine the rate of oral tolerance and identify clinical and laboratory predictors of tolerance development in Thai children who allergic to wheat.

DETAILED DESCRIPTION:
All children in this study were sensitized to wheat. Each patient was clinically evaluated, with focus on wheat allergy by both a detailed medical examination and collection of medical history. Blood sample was taken for baseline determination of ImmunoglobulinE antibodies to wheat and to omega-5-gliadin. The oral wheat challenge were performed in all study subjects to identify a case of wheat outgrowing. The primary outcome was the development of oral tolerance to wheat. Oral wheat challenge were generally performed at least every 1 years if the child did not have an interval history of symptoms with unintentional exposure.

ELIGIBILITY:
Inclusion Criteria:

* children 1 to 15 years
* History of IgE-mediated wheat allergy

Exclusion Criteria:

* Parents refused to sign the consent
* Patient has the underlying disease: congenital heart disease, uncontrolled asthma or life-threatening condition.

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2012-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The number of participants who outgrow from wheat allergy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Punchama Pacharn, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj hospital, Bangkoknoi, Bangkok, Thailand